CLINICAL TRIAL: NCT05449847
Title: Plasma Expression Levels of MicroRNA-21 Might Help for Detection of HCV Patients Complicated by Hepatocellular Carcinoma
Brief Title: Plasma MicroRNA for Prediction of Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amr M. El Hammady, Assistant professor of Internal Medicine, Benha University
Other Study IDs: RC 1.7.2021
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — MicroRNAs (MiR) are naturally occurring short, noncoding RNAs that specifically regulate protein expression and its cumulative effects may lead to broad changes to cell systems and architecture. Deregulated expression levels of MiRs may underlie the development of multiple liver pathologies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complicated HCV
  Interventions: Biological: Blood Sampling
- Non Complicated HCV
  Interventions: Biological: Blood Sampling

INTERVENTIONS:
Biological: Blood Sampling — Blood sampling under a complete aseptic conditions

SUMMARY:
100 patients with diagnosed HCV were evaluated by clinical and ultrasound examination and were categorized as uncomplicated HCV (n=22) and complicated HCV (n=78). All patients were evaluated for hepatosteatosis and liver fibrosis using the computerized hepatorenal index, the hepatic steatosis index, aspartate aminotransferase (AST)/platelet count index (APRI) and the Fibrosis-4 (FIB-4) scores. Blood samples were obtained for estimation of serum levels of liver function tests and plasma levels of microRNA 21 and 126.

ELIGIBILITY:
Inclusion Criteria:

* Complicated hepatitis C by HCC
* Complicated hepatitis C by liver cirrhosis
* Complicated hepatitis C by steatohepatitis
* uncomplicated hepatitis C

Exclusion Criteria:

* pre-portal fibrosis secondary to previous bilharzial disease
* pre-portal fibrosis secondary to alcoholic fatty liver
* The presence of hepatic malignancy other than HCC
* decompensated cirrhosis
* hepatorenal failure
* hepatic manifestations of congestive heart failure.

Ages: 31 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Relation between MicroRNA and HCV | 12 months
  The ability of estimation of plasma microRNA 21 and 126 to differentiate between uncomplicated and complicated HCV patients

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university, Banhā, El- Qalyobia, Egypt